CLINICAL TRIAL: NCT07305792
Title: Effect of High Tone Power Therapy on Pain, Range of Motion and Quality of Life in Lumbosacral Radiculopathy Patients
Brief Title: High Tone Power Therapy on Lumbosacral Radiculopathy Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Lama Saad El-Din Mahmoud, Assistant Professor of Neurology and Neurosurgery Faculty of Physical Therapy October 6 University, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005939
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Radiculopathy Lumbar

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Study group : received the selected physical therapy program in addition to High tone power therapy.
  Interventions: Device: High tone power therapy; Other: selected physical therapy program
- control group (Experimental): received receive a selected physical therapy program only (Therapeutic Ultrasound device, Hot packs and Neurodynamic mobilization for sciatic nerve
  Interventions: Other: selected physical therapy program

INTERVENTIONS:
Device: High tone power therapy — High Tone Power Therapy (HiToP), or High-Frequency External Muscle Stimulation (HTEMS), is an advanced form of electrotherapy that uses medium-frequency sinusoidal currents with simultaneously modulated amplitude and frequency to treat various conditions, especially neurological symptoms and pain
  Arms: study group
Other: selected physical therapy program — selected physical therapy program including (Therapeutic Ultrasound device, Hot packs and Neurodynamic mobilization for sciatic nerve

SUMMARY:
to investigate the effect of High Tone Power Therapy on Pain, Range of Motion and Quality of Life in Lumbosacral Radiculopathy Patients

DETAILED DESCRIPTION:
BACKGROUND: Lumbosacral radiculopathy is a disorder that causes pain in the lower back and hip, as radicular pain is commonly caused by the compression of lumbar spinal nerve roots. High-tone therapy represents a novel form of electrotherapy distinguished from traditional methods by its dynamic modulation of frequency and amplitude. This innovative approach delivers increased energy levels to tissues. Therefore, there has been significant interest in utilizing high-tone therapy for treating various disorders HYPOTHESES: It will be hypothesized that there will be no statically Effect of High Tone Power Therapy on Pain, Range of Motion and Quality of Life in Lumbosacral Radiculopathy Patients RESEARCH QUESTION: Is there an Effect of High Tone Power Therapy on Pain, Range of Motion and Quality of Life in Lumbosacral Radiculopathy Patients

ELIGIBILITY:
Inclusion Criteria:

* Their ages range from 35 to 50 years.
* Both sex.
* Back pain for more than six months; radiating unilaterally down to one lower limb over the dermatomal distributions of L4-L5, L5-S1 nerve roots.
* Radiological confirmation of disc herniation or protrusion at L4-5 or L5-S1 levels by MRI.
* Symptom duration of at least 4 weeks and not more than 6 months.
* Positive Straight Leg Raise test
* Body mass index (18.5 - 24.99Kg/m2).

Exclusion criteria

* Red flags: spinal tumors, cauda equina syndrome, spinal fractures, osteoporosis, infection.
* Bilateral symptoms.
* Spondylolisthesis, spondylitis, spinal canal stenosis.
* Previous lumbopelvic or hip surgery or injection.
* Any hip structural abnormality such as malformations, impingements and degeneration.
* Postural deviations such as scoliosis, kyphosis and lateral shift.
* Fibromyalgia.
* Pregnancy and Gynecological problems.
* Systemic inflammatory conditions (e.g., rheumatoid arthritis and ankylosing spondylitis)
* Uncontrolled chronic conditions (e.g., diabetes mellitus with neuropathy and severe cardiovascular disease)

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain Pressure Threshold Algometer | four weeks
  An algometer is a device used with pressure algometry to measure the pain pressure threshold (PPT), which is the point at which a steadily increasing, non-painful pressure stimulus is perceived as painful.
Back range of motion (BROM) goniometer device | four weeks
  is a specialized instrument, often using inclinometers and magnets, that provides accurate and repeatable measurements of spinal movements such as flexion, extension, rotation, and lateral side bend
The RAND 36-Item Health Survey (Version 1.0) (SF-36) questionnaires, | four weeks
  The RAND 36-Item Health Survey, also known as the SF-36, is a 36-item questionnaire developed by the RAND Corporation to measure health-related quality of life across eight domains: physical functioning, bodily pain, role limitations (due to physical or emotional problems), social functioning, emotional well-being, vitality (energy/fatigue), and general health. It also includes an additional item to assess self-perceived health changes over time.

SECONDARY OUTCOMES:
Visual analogue scale for pain (VAS-P) | four weeks
  The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. VAS has been widely used in diverse adult populations for example; those with rheumatic diseases, patients with chronic pain Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Lama Saad ED Mahmoud, Principal Investigator — October 6 University
Locations (1):
- October 6 University, Giza, El-Sheikh Zayed City Giza 1133 Egypt, Egypt